CLINICAL TRIAL: NCT03523637
Title: Interoceptive Exposure as a Treatment Option for Disabling Fear of Pain: a Single Case Series
Brief Title: Interoceptive Exposure as a Treatment Option for Disabling Fear of Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Aleksandra Puchala, Principal Investigator, University of Leeds
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PY18/100386; IRAS Project ID: 226054 (Other: Integrated Research Application System)
Record Dates: First submitted 2018-04-20; First posted 2018-05-14 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Replicated experimental case series, also called replicated single-subject design or replicated single-case research design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pain Education/Interoceptive Exposure (Experimental): This study will evaluate the effects of IE and will briefly comprises of: education session explaining the rationale behind IE practice, teaching of the technique, supervised IE practice and self-monitored home practice twice daily for the period of two weeks.
  Interventions: Behavioral: Interoceptive Exposure

INTERVENTIONS:
Behavioral: Interoceptive Exposure — The intervention Interoceptive Exposure (IE) is an exposure to bodily sensations used in treatment of variety of problems where body sensations are experienced as threatening. This psychological technique is about focusing attention on pain, 'staying with the pain' without trying to escape it.

SUMMARY:
The aim of this study is to investigate the use of Interoceptive Exposure (IE) in treatment of disabling fear of pain using a single-case series design.

DETAILED DESCRIPTION:
The intervention Interoceptive Exposure (IE) is an exposure to bodily sensations used in treatment of variety of problems where body sensations are experienced as threatening. The application of IE is expected to reduce the threat value of pain and subsequently promote recovery. This study will evaluate the effects of IE and will briefly comprises of: education session explaining the rationale behind IE practice, teaching of the technique, supervised IE practice and self-monitored home practice twice daily for the period of two weeks. Depending on the length of baseline (i.e. observation period before the start of intervention) the study will last between 6 and 8 weeks. Daily Diary, a short nine item instrument was designed to measure the pain experience (intensity and interference) and fear of pain on a daily basis. Other, standard outcome measures include: pain related anxiety, pain catastrophising, pain related disability, knowledge about pain and general anxiety and depression. Study participants will be recruited during routine psychology screening assessment at the Pain Clinic at St James' Hospital. This study will recruit from clinical psychology waiting list patients.

ELIGIBILITY:
Inclusion Criteria:

* Presence of chronic pain (i.e. pain present for minimum of 3 months following tissue damage)
* 18 years or older
* Capacity to give informed consent
* Appropriate diagnostic investigations in other specialties as appropriate have been exhausted and first line interventions, like analgesia, have been tried.
* Participant has appropriate expectations regarding psychological treatment, i.e. does not expect injections etc.

Exclusion Criteria:

* Insufficient understanding of English or additional needs which mean the potential participant is unable to complete questionnaires independently. This is because the research project does not have the resources to make significant adaptations to the materials i.e. translation into another language or into Braille.
* Unable to meet the demands of the study (i.e. daily recording of data, daily practice of IE, coming for sessions to St James' Hospital).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2018-03-05 (Actual); Primary Completion 2018-09-30 (Estimated); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Daily Diary | Assessed daily, throughout the duration of the study. Depending on the length of the baseline this will be between 42 and 56 days.
  The Daily Diary is a 9 item questionnaire used for recording daily ratings of pain distress, pain interference and the fear of pain. Items 1-4 use visual analogue scales (VAS) to measure pain distress and interference. Each VAS has two anchors: "not at all distressing" and "extremely distressing" for pain distress questions (Items 1-3) and "does not interfere" and "interferes completely" for pain interference (Item 4), providing a range of scores between 0 and 100. Higher scores indicate greater pain distress and interference. Additionally, there are 5 statements assessing the fear of pain, which participants rate on a 5 point Likert Scale, where the score of 0 equals "not at all" and score of 4 equals "all the time". An example question: "Pain Sensations are terrifying". Total Fear of Pain Score is calculated by adding up scores on items 5 to 9. Higher Scores indicate higher fear of pain, min = 0, max = 20.
Change in Activity levels, i.e. number of steps taken | Assessed daily, throughout the duration of the study. Depending on the length of the baseline this will be between 42 and 56 days.
  This will be measured with an activity monitor NOKIA GO worn by participants on their wrists or attached to their belt.

SECONDARY OUTCOMES:
Pain Catastrophising Scale (PCS: Sullivan, Bishop & Pivik, 1995) | at three time points: assessment (day one), pre-intervention (depending on the length of the baseline 2 weeks, 3 weeks or 4 weeks later) and post-intervention (6, 7 or 8 weeks from the start of the intervention).
  Standardised measure of pain catastrophising. The PCS is a 13 item scale, with each item rated on a 5-point Likert type scale: 0 (Not at all) to 4 (all the time). Sample item: "I worry all the time about whether the pain will end". The PCS is broken into three sub-scales: magnification, rumination, and helplessness. Scores are added up for each sub-scale, a Total Score is achieved by adding up all 13 items. The higher the score, the more catastrophizing thoughts are present. Previous studies have shown a cutoff of more than 30 points to be associated with clinical relevance.
Pain Anxiety Symptoms Scale Short Scale (PASS-20: McCracken & Dhingra, 2002) | at three time points: assessment (day one), pre-intervention (depending on the length of the baseline 2 weeks, 3 weeks or 4 weeks later) and post-intervention (6, 7 or 8 weeks from the start of the intervention).
  The PASS-20 assesses pain specific anxiety symptoms using four components of pain-related anxiety: cognitive, fear, escape avoidance, and physiological. Each of the four sub-scales has five items. All items are rated from 0 (never) to 5 (always). Sample item: "I worry when I am in pain". Scores are added up for each sub-scale, a Total Score is achieved by adding up all 20 items. The higher the score, the more pain anxiety symptoms. Maximum Total Score: 100, Minimum Total Score: 0.
Pain Disability Index (PDI: Pollard, 1984) | at three time points: assessment (day one), pre-intervention (depending on the length of the baseline 2 weeks, 3 weeks or 4 weeks later) and post-intervention (6, 7 or 8 weeks from the start of the intervention).
  This is a brief self-report measure of disability and is designed to measure the extent to which chronic pain interferes with an individual's ability to engage in activities (Pollard, 1981). Respondents rate the degree to which pain interferes with functioning in seven broad areas: family/home responsibilities, recreation, social activity, occupation, sexual behaviour, self-care, and life-support activity on a ten-point scale of 0 (no disability) to 10 (total disability). Sample Item: "Recreation: This disability includes hobbies, sports, and other similar leisure time activities". An overall score (with a possible total of 70) is computed by summing the seven sub-scales, higher scores indicate greater level of pain related disability. Validity and reliability have been established for this measure (Tait, Chibnall and Krause, 1990).
Hospital Anxiety and Depression Scale (HADS: Zigmond & Snaith, 1983) | at three time points: assessment (day one), pre-intervention (depending on the length of the baseline 2 weeks, 3 weeks or 4 weeks later) and post-intervention (6, 7 or 8 weeks from the start of the intervention).
  Standardised questionnaire used in assessing generalised anxiety and depression. The questionnaire comprises seven questions for anxiety and seven questions for depression (total number of items = 14). Each item on the questionnaire is scored from 0 - 3 and this means that a person can score between 0 and 21 for either anxiety or depression. Sample Item: "I feel tense or 'wound up'", response options: "Most of the time" (scored 3 points), "A lot of the time" (Scored 2 points), "From time to time" (Scored 1 point), "Not at all" (Scored 0 points). Although the anxiety and depression questions are interspersed within the questionnaire, they can be added up together (Total Score) or added up within each sub-scale (Depression Total Score and Anxiety Total Score). Higher scores are indicative of more symptoms of Generalised Anxiety and Depression.
Chronic Pain Acceptance Questionnaire (CPAQ: McCracken, Vowles & Eccleston, 2004) | at three time points: assessment (day one), pre-intervention (depending on the length of the baseline 2 weeks, 3 weeks or 4 weeks later) and post-intervention (6, 7 or 8 weeks from the start of the intervention).
  Standardised questionnaire used in assessing the acceptance of pain in chronic pain sufferers. The CPAQ assesses acceptance of pain using two factors: Activity Engagement (participation in daily activities while acknowledging the presence of pain, 11 items) and Pain Willingness (the degree to which pain is allowed in experience without efforts to avoid or control it; 9 items). Sample Item: "My life is going well, even though I have chronic pain". The items on the CPAQ are rated on a 7-point scale from 0 (never true) to 6 (always true). Scoring is done by adding the items for Activity engagement and Pain willingness to obtain a Total Score for each factor. Additionally, a total score of Pain Acceptance is calculated by adding the scores for each factor together. Higher scores indicate higher levels of acceptance. Maximum Total Acceptance Score is 120, Minimum Total Acceptance Score is 0.

CONTACTS AND LOCATIONS:
Locations (1):
- Pain Clinic, Fielding House at St James's Hospital, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No